CLINICAL TRIAL: NCT05588245
Title: A Pragmatic Trial of Integrating Community-based Patient Navigation Into the Continuum of Maternal Care for Black Women in a Safety-Net Health System: Effects on Maternal Health, Health Care, Morbidity, and Mortality
Brief Title: Trial of Community-based Patient Navigation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Anne Lang Dunlop, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004987; R01NR020756-02 (NIH)
Record Dates: First submitted 2022-10-18; First posted 2022-10-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Comparison Group (Standard of Care) (Active Comparator): Participants will receive the standard of care.
  Interventions: Behavioral: Standard of Care
- Intervention Group (Experimental): Participants will receive a community-based patient navigator with 3 prenatal contacts and 5 postpartum contacts; during each contact, the community-based patient navigator will offer health assessment and education, along with group education and social support.
  Interventions: Behavioral: Community-based prenatal/perinatal/postpartum patient navigator

INTERVENTIONS:
Behavioral: Standard of Care — Participants will undergo the same SDoH screener (AHC-Health Related Social Needs Tool) as full intervention participants, which will serve as the basis for a one-time brief session with the clinical research coordinator that will involve review of a 'Resource Guide' that provides a listing of available community resources to meet common social needs. Participants in this arm will also complete other prenatal and postpartum data collection items over the course of the study (with the exception of qualitative interviews).
  Arms: Comparison Group (Standard of Care)
Behavioral: Community-based prenatal/perinatal/postpartum patient navigator — Uses Freeman's principles of navigation to enhance patient access to care (e.g., help patients manage appointments), promote patient self-efficacy (e.g., connect patients to community housing, food, transportation resources), and sustain engagement with the healthcare system (e.g., bridge perinatal and primary care).
  Other Names: PPP-PN
  Arms: Intervention Group

SUMMARY:
This study will test the effectiveness of a community-based patient navigator intervention from mid-pregnancy through 12 month postpartum for a high-risk population of medically underserved women. The RCT will enroll 540 pregnant women before 20 weeks of pregnancy and randomly allocate them into two different study arms from the time of prenatal enrollment through 12 months postpartum. If found to be effective, the community-based patient navigator intervention can be implemented as a standard of care at Grady and other provider practices serving high-risk women to improve maternal health outcomes and reduce racial disparities.

DETAILED DESCRIPTION:
Severe maternal morbidities (SMM) are outcomes of labor and delivery that result in serious effects on short- or long-term health. Many SMM represent "near miss" events for maternal deaths. In Georgia, Black women experience SMM at a rate far higher than women of other races and ethnicities. Equity-centered models of care - such as embedding patient navigators into the maternity care continuum - offer promise for improving maternal health through meeting the social needs, lowering stress, and promoting access to and utilization of care for those giving birth. To date, however, research about maternity care navigation's effectiveness and needed inputs for its adoption into clinical care are lacking. To fill this research gap, the investigators propose to complete a pragmatic randomized controlled trial (RCT) of integrating community-based patient navigators into maternal care of Black women being cared for through Grady Health System (a safety net health system in Atlanta). The RCT will enroll 540 pregnant women before 20 weeks of pregnancy and randomly allocate them into two different study arms from the time of prenatal enrollment through 12 months postpartum. The first arm (the comparison group) will receive the standard of care. The second arm (the intervention group) will receive a community-based patient navigator with 3 prenatal contacts and 5 postpartum contacts; during each contact, the community-based patient navigator will offer health assessment and education, along with group education and social support. For participants in both arms, the researchers will collect data on patient-level measures upon enrollment (<20 weeks' of pregnancy), at 6-8 weeks postpartum, and at 12 months postpartum; data collection will involve questionnaires, review of case logs and review of medical records. Measures of effectiveness will include the number of SMM and maternal death events per woman (primary outcome). To evaluate how the intervention might reduce primary outcomes, questionnaires will also assess measures of unmet need, stress and depressive symptoms, attendance of prenatal and postpartum care. Embedded process evaluation will assess the number and content of navigation encounters in which the woman participates and the acceptability of the intervention from patient and provider perspectives.

Written informed consent will be obtained as a criterion for participation. All participants will be compensated for their time. Confidentiality will be maintained on several levels including training of investigators and staff, restrictions on data access, and use of HIPPA-compliant data storage procedures. Data will be stripped of identifiers before analysis and destroyed when no longer needed.

This study will be among the first to test the effectiveness of a community-based patient navigator intervention from mid-pregnancy through 12 month postpartum for a high-risk population of medically underserved women. If found to be effective, the community-based patient navigator intervention can be implemented as a standard of care at Grady and other provider practices serving high-risk women to improve maternal health outcomes and reduce racial disparities.

ELIGIBILITY:
Inclusion Criteria:

* A pregnant woman or individual (inclusive of all gender identities) who is Black and English-speaking (by self-report),
* ≥18 years of age who is capable of consenting for oneself and who presents for prenatal care with a singleton pregnancy ≤ 20 weeks gestation (confirmed by medical record),
* covered by Medicaid
* for whom the AHC-Health Related Social Needs Tool (administered as part of standard clinical care for prenatal patients) identifies ≥1 unmet social needs
* expectation to receive prenatal care and deliver at Grady and be available through 12-months postpartum to assure opportunity for exposure to the intervention, process, and outcome measure ascertainment.

Exclusion Criteria:

* The intent to transfer care to a health system outside of metro Atlanta
* incarceration, which would interfere with intervention provision and outcome ascertainment
* adults unable to give consent
* individuals who are not yet adults
* prisoners
* cognitively impaired individuals with impaired decision-making capacity
* individuals who are not able to clearly understand and speak English (as the PPP-PN intervention is only available in English at this time)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in number of SMM and maternal death events | Baseline, 12 months postpartum
  This is a count measure that reflects the total number of SMM and/or death events during the delivery admission through 12-months of delivery according to the presence/absence of the 21 SMM indicator diagnosis codes (as published by the Centers for Disease Control and Prevention) and/or a death event documented in the EPIC electronic medical record.

SECONDARY OUTCOMES:
Change in number of post-delivery maternal morbidity (non-SMM) events | Baseline, 12 months postpartum
  This is a count measure that reflects the total number of specific non-SMM maternal morbidities according to the presence/absence of ICD-10 diagnostic codes for postpartum hemorrhage without transfusion, hypertensive disorders, endometrial infection, venous thrombosis, depression or anxiety, substance use disorder for an emergency department visit or re-hospitalization event in the EPIC electronic medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Dunlop, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data related to the primary and secondary endpoints will be shared, including severe maternal morbidity (SMM) and death events, health care utilization data, health care quality data (receipt of guideline concordant care), and patient-reported outcomes (unmet social needs, emotional support, quality of life, perceived stress and depression, substance use, perceptions of care, satisfaction with care)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available in the final year of the study (Year 5, anticipated starting September 2026) when all data collection is complete and will be available thereafter.
Access Criteria: Consistent with the NIH Data Sharing Policy, the investigators will make the de-identified data and associated documentation available to users under a data-sharing agreement. To gain access to study data, anyone not part of the original research protocol will submit a Data Analysis Request Form, which requires elucidation of the specific data requested along with a statement that the investigator must provide: 1) a commitment to using the data only for research purposes and not to identify any individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed.